CLINICAL TRIAL: NCT06675370
Title: Validity and Reliability of the Glittre Activities of Daily Living Test for Assessing Functional Status in Individuals With Chronic Low Back Pain
Brief Title: The Glittre Activities of Daily Living Test in Chronic Low Back Pain
Status: Completed | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-14/121
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2024-11

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Indıviduals with chronic low back pain

SUMMARY:
The aim of our study is to investigate the validity and reliability of the Glittre activities of daily living test in individuals with chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic low back pain
* Chronic low back pain for at least the last 3 months
* Being aged 18-65
* Voluntary participation in the study

Exclusion Criteria:

* Having orthopedic or neurological impairments
* History of surgery due to chronic low back pain in the last 6 months
* Being pregnant
* Participating in regular physical activity in the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals with chronic low back pain who are being followed up at the Department of Physical Medicine and Rehabilitation at Kirsehir Ahi Evran University will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2024-11-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
Daily living activities | 20 minutes
  It will be evaluated with the Glittre activities of daily living test
Exercise capacity | 10 minutes
  It will be evaluated with 6 minute walk test.

SECONDARY OUTCOMES:
Musle function | 1 minute
  It will be assessed with a one-minute sit-stand test.
Functional mobility | 1 minute
  This will be evaluated with a timed up and go test.
Disability level | 5 minutes
  It will be assessed with Oswestry Disability Index. High scores on the scale indicate the presence and severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Firat, Principal Investigator — Kirsehir Ahi Evran University; Basak Kavalci Kol, Study Chair — Kirsehir Ahi Evran University; Figen Tuncay, Study Chair — Kirsehir Ahi Evran University
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)